CLINICAL TRIAL: NCT02067000
Title: Validation of the Patient Perception Questionnaire
Brief Title: Patient Perception Questionnaire Validation
Status: Completed | Type: Observational
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CIA-44
Record Dates: First submitted 2013-09-12; First posted 2014-02-20 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obstructive Sleep Apnea
  Interventions: Behavioral: Obstructive Sleep Apnea

INTERVENTIONS:
Behavioral: Obstructive Sleep Apnea — Questionnaire about CPAP perceptions

SUMMARY:
Validation of the patient perception questionnaire relating to CPAP use

DETAILED DESCRIPTION:
This research is designed to validate a questionnaire which aims to predict patient adherence to CPAP, therefore enabling the healthcare provider to better target initiatives to improve adherence.

ELIGIBILITY:
Inclusion Criteria:

* Mild-severe OSA patients
* Over 18
* Naive to CPAP
* Fluent english

Exclusion Criteria:

* Comorbidities
* Other sleep disorders
* Inability to tolerate CPAP
* Shift worker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OSA patients
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Powell, Principal Investigator — Clayton Sleep Institute
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obstructive Sleep Apnea
Started | 217
Completed | 167
Not Completed | 50

BASELINE CHARACTERISTICS:
Arm/Group | Obstructive Sleep Apnea
Number analyzed (Participants) | 217
Age, Continuous [Mean (Full Range); unit: Years] | 54.1 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 170
  Other | 47
Region of Enrollment [Number; unit: participants]
  United States | 217

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Association of the Participants Baseline PPQ (Patient Perception Questionnaire) Responses to Predict Adherence to CPAP Treatment at 90 Days.
Description: The PPQ is a custom questionnaire including 10 questions evaluating perceptions of OSA and CPAP treatment. Each question is derived from models of psychology such as self-regulatory ability and social support. Q1 ranges from 0-10, with 10 indicating OSA negatively impacts life. Q2 ranges from 0-10, with 10 indicating belief that OSA will last forever. Q3 ranges from 0-10, with 10 indicating that CPAP is extremely necessary to control OSA. Q4 ranges from 1-10, with 10 indicating no intention of using CPAP at all. Q5 ranges from 1-10, with 10 indicating presence of a highly supportive spouse. Q6 ranges from 1-10, with 10 indicating benefit of CPAP is well understood. Q7 ranges from 0-10, with 10 indicating extreme concern about using CPAP. Q8 ranges from 1-10, with 10 indicating high confidence with using CPAP. Q9 ranges from 1-10, with 10 indicating high perception that CPAP will help treat OSA. Q10 ranges from 1-10, with 10 indicating spouses negative attitude toward CPAP use.
Time Frame: Baseline and 90 days
Measure: Number; unit: r value
Arm/Group | Obstructive Sleep Apnea
Number analyzed (Participants) | 167
r value
  Q1 | .04
  Q2 | .14
  Q3 | .10
  Q4 | .13
  Q5 | .25
  Q6 | .01
  Q7 | .29
  Q8 | .16
  Q9 | .12
  Q10 | .19

2. Secondary Outcome: Adherence to CPAP Treatment
Description: An assessment of participants adherence to CPAP treatment after 90 days. Data was extracted from CPAP device compliance reports.Adherence was defined as use for 4 hours or more per night for 70% of nights in each report period at 14, 60 and 90 days.
Time Frame: 14 Days, 60 Days, 90 Days
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Obstructive Sleep Apnea
Number analyzed (Participants) | 161
Minutes
  14 Days | 335 (118)
  60 Days | 322 (118)
  90 Days | 317 (119)

3. Secondary Outcome: Reliability of Patient Perception Questionnaire
Description: To determine the stability/consistency (reliability) of the PPQ at three time points during the first 90 days of CPAP treatment usage. At each of these time points, the exact same PPQ as described in the Primary Outcome Measure was re-administered to determine whether the scores remained consistent over time. The answer responses described in the Primary Outcome measure also remain the same. Total PPQ was calculated as an average of the 10 questions. Total score ranges from 0-10 with higher scores indicating a worse outcome.
Time Frame: 14 days, 60 days, 90 days
Population: Due to missing or incomplete data and drop outs, only participants who had completed all 10 questions of the PPQ were included in the analysis for each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obstructive Sleep Apnea
Number analyzed (Participants) | 167
units on a scale
  14 days: number analyzed (Participants) | 162
  14 days | 6.43 (0.99)
  60 days: number analyzed (Participants) | 58
  60 days | 6.35 (0.92)
  90 days: number analyzed (Participants) | 36
  90 days | 6.06 (1.14)

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Obstructive Sleep Apnea
All-Cause Mortality (participants affected / at risk) | 0/217
Serious Adverse Events (participants affected / at risk) | 0/217
Other Adverse Events (participants affected / at risk) | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No